CLINICAL TRIAL: NCT06238791
Title: Static Plantar Pressure Distribution and Presence of Foot Deformities in Patients With Lipedema and Chronic Venous Disease
Brief Title: Plantar Pressure Analysis and Foot Biomechanics in Lipedema and Chronic Venous Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zilan Bazancir Apaydın, Asst. Prof., Hacettepe University
Other Study IDs: 2023 - 1151
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Chronic Venous Insufficiency; Lipedema
Keywords: Foot deformity; venous insufficiency; pressure; Lipedema
MeSH Terms: conditions — Lipedema; Foot Deformities; Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic venous disease group
  Interventions: Other: Presence of foot deformity, ankle range of motion, foot posture, local tissue water percentage, and foot pressure distribution will be evaluated in patients with chronic venous disease.
- Chronic venous disease and lipedema group
  Interventions: Other: Presence of foot deformity, ankle range of motion, foot posture, local tissue water percentage, and foot pressure distribution will be evaluated in patients with chronic venous disease.

INTERVENTIONS:
Other: Presence of foot deformity, ankle range of motion, foot posture, local tissue water percentage, and foot pressure distribution will be evaluated in patients with chronic venous disease. — Presence of foot deformity, ankle range of motion, foot posture, local tissue water percentage, and foot pressure distribution will be evaluated in patients with chronic venous disease and lipedema.

SUMMARY:
Chronic venous disease (CVD) are common vascular pathology characterized by a wide spectrum of clinical manifestations occurring with symptoms and/or signs that vary in type and severity. The pathophysiological mechanisms of CVD start from the development of venous hypertension, leading to endothelial dysfunction and venous wall dilatation. Lipedema is subcutaneous adipose tissue disorder characterized by enlargement of both lower extremities. Previous studies showed that foot deformities such as pes planus or cavus are at a high prevalence in CVD patients, and the authors indicated that foot disorders are an important risk factor that negatively affects venous disease. To the best of our knowledge, there is only one study investigating plantar arch abnormalities in lipedema patients based on clinical observation. Therefore, the study aimed to investigate plantar foot distribution and foot deformity in patients with CVD and lipedema.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with CVD or CVD combined with lipedema,
* The clinic (C) score of clinical, etiological, anatomical, pathophysiological (CEAP) classification was C1, C2 or C3 (C1: telangiectasia-reticular vein; C2: varicose vein; C3: edema)

Exclusion Criteria:

* C4, C5 or C6 (presence of skin changes or ulcer) in C score of CEAP classification
* undergone lower extremity orthopedic surgery within the last year,
* have peripheral artery disease
* patients who could not mobilize independently

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were divided into two groups: Patients with only CVD and patients with CVD accompanied lipedema.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
The presence of foot deformity | baseline of study
  The presence of foot deformity including hallux valgus, hallux limitus or rigidus, pes planus, pes cavus, toe deformities will be evaluated by inspection. In the presence of hallux valgus, its stage will be evaluated by measuring the angle using a universal goniometer, and in the presence of pes planus, the severity of pes planus will be determined by performing the navicular drop test.
Plantar pressure distribution | baseline of study
  Plantar pressure distribution (PPD) will be evaluated with EsCoSCAN® (EsCo Orthopädie Service GmbH, Germany) pedobarography. The plantar pressure in both feet will be evaluated with the force platform while standing, and the average pressure distribution percentage for each foot will be recorded.

SECONDARY OUTCOMES:
Ankle range of motion | baseline of study
  Ankle dorsi- and plantar-flexion range of motion will be measured using a universal goniometer.
Foot posture | baseline of study
  The foot posture will be evaluated with the Foot Posture Index.
Local tissue water percentage | baseline of study
  Local tissue water percentages will be evaluated with the Moisturemeter-d compact (MMDc, Delfin Technologies, Kuopio, Finland) device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uhl JF, Chahim M, Allaert FA. Static foot disorders: a major risk factor for chronic venous disease? Phlebology. 2012 Feb;27(1):13-8. doi: 10.1258/phleb.2011.010060. Epub 2011 Jul 4. PMID 21727156
- [Result] Forner-Cordero I, Szolnoky G, Forner-Cordero A, Kemeny L. Lipedema: an overview of its clinical manifestations, diagnosis and treatment of the disproportional fatty deposition syndrome - systematic review. Clin Obes. 2012 Jun;2(3-4):86-95. doi: 10.1111/j.1758-8111.2012.00045.x. Epub 2012 Aug 3. PMID 25586162